CLINICAL TRIAL: NCT05221190
Title: Comparative Evaluation of the Effectiveness of Buccal Infiltration Anesthesia Versus Inferior Alveolar Nerve Block Anesthesia for the Extraction of Primary Mandibular Molars: A Randomized Controlled Study
Brief Title: Buccal Infiltration Anesthesia Versus Inferior Alveolar Nerve Block Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa aly fouad elchaghaby, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anesthetic techniques
Record Dates: First submitted 2022-01-03; First posted 2022-02-02 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single buccal infiltration of articaine anesthesia (Experimental): The local anesthetic solution will be administered using single buccal infiltration with articaine anesthesia.
  Interventions: Procedure: Single buccal infiltration
- Inferior alveolar nerve block of lidocaine anesthesia (Active Comparator): The anesthetic solution will be administered using inferior alveolar nerve block with lidocaine anesthesia.
  Interventions: Procedure: Inferior alveolar nerve block

INTERVENTIONS:
Procedure: Single buccal infiltration — injecting local anaesthetic solution into the soft tissues of the buccal sulcus adjacent to the target tooth.
  Other Names: Articaine buccal infiltration
  Arms: Single buccal infiltration of articaine anesthesia
Procedure: Inferior alveolar nerve block — Injection of local anesthetic solution into the pterygomandibular space to access the inferior alveolar nerve before it enters the mandible.
  Other Names: Lidocaine nerve block
  Arms: Inferior alveolar nerve block of lidocaine anesthesia

SUMMARY:
This study aims to evaluate the effectiveness of single buccal local infiltration when compared to buccal local infiltration with intrapapillary infiltration and inferior alveolar nerve block anesthesia in primary mandibular molar extractions.

DETAILED DESCRIPTION:
Effective pain control is essential in providing children with successful dental treatment. Without it, negative experiences may result in anxiety and fear-related behaviors towards subsequent dental treatment. Local anesthesia is the cornerstone of pain control in dentistry. Choosing the right local anesthetic technique is of special significance .

The inferior alveolar nerve block (IANB) is a common practice for anesthetizing mandibular molars and/or premolars on one side of the jaw. It is achieved by depositing local anesthetic solution at the entrance to the mandibular canal, which inhibits the transmission of action potentials along the inferior alveolar nerve.

Administering an IANB can be technique sensitive and failure rates are reported to be up to 20%, due to anatomical variations in the position of the mandibular foramen and accessory innervations. This effect may be compounded for those who are not used to anesthetizing children .

However, Supraperiosteal infiltration has the advantages of easier administration when compared to block anesthesia, shorter anesthetic duration, and generally does not anesthetize the lips .

An ideal local anesthetic should provide maximum efficacy, through a minimal number of injections, using techniques that provide the least discomfort, causing negligible adverse effects .

ELIGIBILITY:
Inclusion Criteria:

* Badly decayed primary mandibular molars indicated for extraction with not less than half of the root length present.
* Children ranging in age from 5-8 years

Exclusion Criteria:

.Allergies to local anesthetics.

* History of significant medical conditions.
* Children under any medications.
* Presence of abscess, sinus opening.
* Uncooperative children without access to or with difficulty accessing dental care.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Assessment of intraoperative pain | through treatment completion, an average of 1 hour
  Wong Baker Faces Pain Rating Scale consists of a set of cartoon faces with varying facial expressions ranging from a smile/laughter to tears with numerical value from 0 to 5 where where zero indicates no pain and 5 indicate severe pain

SECONDARY OUTCOMES:
intraoperative pain | through treatment completion, an average of 1 hour
  Faces, Legs, Activity, Cry, and Consolability scale with score from 0 to 10 where zero indicates no pain and 10 indicate severe pain
The onset of the anesthetic effect | up to 24 hours
  stopwatch
duration of the anesthetic effect | up to 24 hours
  stopwatch

CONTACTS AND LOCATIONS:
Overall Officials: marwa m elchaghaby, phd, Principal Investigator — marwaaly2003@yahoo.com
Locations (1):
- Cairo university, Cairo, Egypt